CLINICAL TRIAL: NCT04777383
Title: A Non-randomized Experimental Study of Optically Registered Pharmacodynamic Responses During Iontophoresis of Vasoactive Substances to the Skin of Healthy Volunteers
Brief Title: The Effects of Iontophoresed Vasoactive Drugs on Cutaneus Blood Flow
Acronym: Jonto01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, Principal investigator, University Hospital, Linkoeping
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-004624-11
Record Dates: First submitted 2021-02-22; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Diseases; Vascular Diseases
Keywords: iontophoresis; pharmacology; tissue viability imaging; multi-exposure laser speckle contrast imaging
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases | interventions — Acetylcholine; Norepinephrine; Phenylephrine; Atropine; Neostigmine

STUDY DESIGN:
Intervention Model Description: Iontophoresis of vasoactive substances in 5 different concentrations. Each concentration is administrated 3 times to the same localisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vascular effects of iontophoresed vasoactive substances (Experimental): Iontophoretically administered vasoactive substances in five concentrations (1%,0.1%,0.01%,0.001%, 0.0001%) dissolved in sterile water. Each concentration of the drug is separately administered using a electrical charge of 12 millicoulomb (mC) (600 seconds x 0.02 milliampere) for 3 repeated pulses (total electrical charge 36 mC). Each iontophoresis pulse is separated by a 30 minute wash-out period.
  Vasoactive substances:
  * Miochol-E (Acetylcholine),10 mg/ml, Bausch & Lomb
  * Methacholine chloride, 100 mg/ml, APL
  * Norepinephrine, 1 mg/ml, Pfizer
  * Phenylephrine, 10 mg/ml, Unimedic
  * Atropine, 10 mg/ml, Bausch & Lomb
  * Neostigmine, 2.5 mg/ml, Unimedic Pharma
  * Sterile water, 100 ml, Braun
  Interventions: Drug: Acetylcholine; Drug: Norepinephrine; Drug: Phenylephrine; Drug: Atropine; Drug: Neostigmine; Drug: Sterile water

INTERVENTIONS:
Drug: Acetylcholine — Iontophoretic administration of 5 different concentrations of acetylcholine
  Other Names: Miochol-E, 10mg/ml, Bausch and Lomb
Drug: Norepinephrine — Iontophoretic administration of 5 different concentrations of norepinephrine
  Other Names: Norepinephrine, 1 mg/ml, Pfizer
Drug: Phenylephrine — Iontophoretic administration of 5 different concentrations of phenylephrine
  Other Names: Phenylephrine, 10 mg/ml, Unimedic
Drug: Atropine — Iontophoretic administration of 5 different concentrations of atropine
  Other Names: Atropine, 10 mg/ml, Bausch & Lomb
Drug: Neostigmine — Iontophoretic administration of 5 different concentrations of neostigmine
  Other Names: Neostigmine, 2.5 mg/ml, Unimedic Pharma
Drug: Sterile water — Iontophoretic administration of sterile water
  Other Names: Sterile water, 100 ml, Braun

SUMMARY:
Many acute and chronical medical conditions, such as, shock, sepsis, diabetes, hypertonia, and cardiovascular disease are associated with a perturbated or lost ability of regulating the diameter of the blood vessels. These changes in regulatory function can be seen especially in the smaller vessels in the body. It is therefore clinically relevant to develop investigation models that can detect and quantify such changes at an early stage.

Historically, basic vascular function was investigated by mounting a section of a blood vessel on a tension sensor, submerging it in a temperature controlled and buffered solution to which vasoactive substances were added. This in vitro model has contributed substantially to our current knowledge of vascular pharmacology and function. However, using this method means that the vessel is removed from its natural environment and, hence no longer influenced by systemic or local mediators for controlling vessel diameter.

The present study aims to investigate the local changes in blood flow and concentration of red blood cells of the superficial vessels in the skin of the forearm of healthy volunteers in response to various vasoactive substances. The purpose is to better understand how the regulation of diameter works in and to find a model that can give an early warning to when it does not function optimally.

The vasoactive substances will be delivered through the skin to the vascular bed by a non-invasive method called iontophoresis. An electrode chamber containing a solution of the substance to be studied is placed on the subject's skin by double adhesive tape. The chamber comes with a transparent lid that prevents leakage and enables supervision of the effect on the underlying vasculature. When a voltage is applied the charged drug molecules begin to move through the skin and interact with the vessels. In the present study, a total electrical dose of 12 millicoulomb (mC) is going to be used (600 seconds x 0.02 milliampere).

The effect of the applied drug is measured using two non-contact, optical measurement techniques.

A better understanding of the pharmacology and regulation of blood vessels may lead to the developement of techniques that allow earlier detection of perturbations in vessel regulation and the onset of preventive medical treatment.

DETAILED DESCRIPTION:
A non-randomised study to investigate how 6 different vasoactive substances administrated in 5 different concentrations, and with repeated administration affect the cutaneous superficial vessels. The primary aim is to investigate dose-response mechanisms by use of two non-invasive optical measurement technologies.

The substances are administrated by iontophoresis using a protocol with a current of 0.02 mA for 600 seconds, at a total electrical charge of 12 mC. Each drug is diluted using sterile water into five concentration (1%, 0.1%, 0.01%, 0.001% and 0.0001%). In the sixth chamber only sterile water will be administrated.

An electrode chamber per concentration is attached to the skin of each subject's forearm and each concentration is administrated three times.

Only one substance at a time will be administrated.

The substances used are:

* Acetylcholine - vasodilator (Miochol-E, 10mg/ml, Bausch and Lomb)
* Noradrenaline - vasoconstrictor (Noradrenaline, 10mg/ml, Pfizer)
* Phenylephrine - vasoconstrictor (Phenylephrine, 10mg/ml, Unimedic)
* Atropine - anticholinergic (Atropine, 10mg/ml, Bausch and Lomb)
* Neostigmine - acetylcholineesterase inhibitor (Neostigmine, 10mg/ml, Unimedic Pharma)
* Dilutor: sterile water (Sterile water, 100 ml, Braun)

Iontophoresis protocol: 0.02 mA x 600 seconds x 3 repetitions per drug concentration and localization. Each iontophoretic pulse is preceded by a baseline registration and followed by a 30 minutes wash-out/recovery period.

Vascular effects are continuously, non-invasively and indirectly measured using tissue viability imaging (TiVi, cross-polarized diffuse reflectance spectroscopy) and multi-exposure laser speckle contrast imaging (MELSCI). The optical measurement modalities are placed at a distance of approximately 30 cm above the skin surface so that the vascular responses can be measured in three electrode chambers simultaneously for the duration of the test (120 minutes).

TiVi settings - 1 image/minute at 6000 x 4000 pixels MELSCI settings - 15.6 frames/second at 1024 x 1000 pixels

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No ongoing medication
* No skin disease or other skin afflictions
* Informed, voluntary participation

Exclusion Criteria:

* Ongoing medication (contraceptives excluded)
* Hypertonia, skin disease or skin afflictions, cardiovascular disease, pregnancy
* Damaged skin, bruises, scar tissue or tattoos on the skin of the forearms
* Smoking (6 months prior to study onset, or more than 100 cigarettes in life)
* Snus (6 months prior to study onset)
* Use of nicotine products (gum, patch, et cetera) 6 months prior to study onset
* Blood pressure above 140/90
* Coffee, tea, alcohol or strenuous physical activity on the day of the study
* Not fasting for 2 hours prior onset of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Locally induced changes in red blood cell concentration and movement due to iontophoresis of vasoactive substances. | Measured prior the onset of iontophoresis (baseline), then continuously for the duration of the iontophoretic pulse (10 minutes) and for the 30 minute wash-out period following each iontophoretic pulse.
  Optically derived arbitrary values that correlate to the concentration and movement of red blood cells in the vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wilhelms, Phd, Principal Investigator — Linkoeping University
Locations (1):
- University Hospital Linköping, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Henricson J, Sjoberg F, Iredahl F, Stromberg T, Wilhelms D. In vivo dose-response analysis to acetylcholine: pharmacodynamic assessment by polarized reflectance spectroscopy. Sci Rep. 2022 Apr 21;12(1):6594. doi: 10.1038/s41598-022-10617-x. PMID 35449189